CLINICAL TRIAL: NCT06589908
Title: Evaluation of the Use of RELAX Glasses on Anxiety of Patients Undergoing Dental Extraction > 2 Teeth, Under Local Anesthesia, Compared With Those Not Using Glasses
Acronym: BRIGAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Valenciennes (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-02-02
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2024-09

CONDITIONS: Surgery
Keywords: audiovisual sedation; anxiety; dental extraction; local anesthesia
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group with RELAX glasses (Experimental): Behavioral : RELAX glasses Glasses which are a solution of audiovisual sedation by positive distraction for hospital medical use
  Interventions: Behavioral: RELAX glasses
- Group without RELAX glasses (No Intervention)

INTERVENTIONS:
Behavioral: RELAX glasses — Glasses which are a solution of audiovisual sedation by positiv distraction for hospital medical use
  Arms: Group with RELAX glasses

SUMMARY:
The vast majority of tooth extraction surgery is performed under local anaesthetic, and can be a source of anxiety. In their 2015 article, Appukuttan et al studied the anxiety felt by 1148 patients prior to tooth extraction, and reported up to 82% of patients anxious before a procedure.

In 2020, Yamashita et al demonstrated the value of virtual reality in reducing patient anxiety during the extraction of three impacted mandibular molars, with no clear effect on the pain felt by the patient.

The use of a virtual reality headset has been shown to reduce anxiety in dental surgery or in hand surgery under local anesthesia with the WALANT technique. On the other hand, virtual reality and the use of 3D can cause discomfort and side effects such as nausea and dizziness. Audiovisual distraction is also known to be effective in reducing pain and anxiety in patients, with fewer side effects.

The investigators have therefore chosen to use RELAX® eyewear. They wish to study its effect on anxiety, pain and overall patient and surgeon satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing dental extraction > 2 teeth under local anesthesia;
* Over 14 years of age on the day of inclusion;
* Patient with written consent or additional parental consent for minors;
* Socially insured patient;
* Patient willing to comply with all study procedures and duration.

Exclusion Criteria:

* Medical history contraindicating RELAX glasses
* Known and current abuse of alcohol and/or illicit drugs that may interfere with patient safety and/or compliance;
* Any condition that would render the patient unfit for the study: current presence of cognitive disorders (MMS < 15), severe psychiatric disorders (bipolar disorders, psychotic disorders according to DSM-V classification);
* Major anxiety requiring preoperative anxiolytics;
* Patient under court protection;
* Patient participating in another study;
* Patient's refusal to use glasses;
* Visually impaired or blind patient.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in visual analogue scale anxiety scores after tooth extraction | In the 5 minutes after the end of surgery
  The visual analogue anxiety scale from 0 to 10, with meaning no anxiety and 10 very high anxiety

SECONDARY OUTCOMES:
Overall satisfaction between the group using RELAX glasses and the group following the usual course (without RELAX glasses) measured by a visual analogue scale | Immediative postoperative
  The visual analogue satisfaction scale ranges from 0 to 10, with 0 eaning unsatisfaction and 10indicating very high satisfaction
Variation in pain between entering and leaving the surgical technical platform between the 2 arms using a visual analogue scale | In the 5 minutes after the end of surgery
  The visual analogue pain scal range from 0 to 10, with 0 meaning non pain and 10 very high pain
Rate of patients receiving at least one analgesic | After local anesthesia
Surgeon's satisfaction with the feasibility of the procedure in a patient wearing RELAX glasses filling in a self-assessment questionnaire | Immediative postoperative
  Self-assessment questionnaire consists of 2 questions :
  Assessment of the severity of the operation on a scale of 0 to 10. 0 indicates no severity and 10 extreme severity.
  Assessment of patient compliance on a scale from 0 to 10. 0 indicating that the patient was completely compliant and 10 indicating absolutely non-compliant.
Pre-existing anxiety, only in patients receiving RELAX glasses, measured with the STAI-YB score | 7 days (+/-3 days) after surgery
  Only in patients receiving RELAX glasses : if the STAY-IB score is higher than 65, the patient is considered to have pre-existing anxiety
Evaluation of the impact of patient agitation on the operative procedure by filling in a self-assessment questionnaire after each operative procedure. | Immediative postoperative
  The questionnary consists of 5 statements. The surgeon must tick only one of them (it's not a scale)
  * the patient was not agitated
  * The patient was agitated, but this had no impact on the surgical procedure
  * Patient agitation caused a change in the surgical procedure
  * Patient agitation was the cause of a temporary suspension of the surgical procedure
  * The patient's agitation is too great to consider continuing the procedure under local anaesthetic.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Valenciennes, Valenciennes, France, France

IPD SHARING:
Plan to Share IPD: No